CLINICAL TRIAL: NCT03068494
Title: Multicenter, Retrospective Korean Coronary Bifurcation Stenting (COBIS) Registry III
Brief Title: Korean Coronary Bifurcation Stenting (COBIS) Registry III
Acronym: COBIS III
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Other Study IDs: 2016-12-136
Record Dates: First submitted 2017-02-27; First posted 2017-03-01 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Coronary Bifurcation Lesion
Keywords: Coronary Bifurcation Lesion; 2nd generation drug-eluting stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Bifurcation Lesion

SUMMARY:
The COBIS III registry is a multi-center, real-world registry of 2nd generation drug-eluting stenting in coronary bifurcation lesions in South Korea. From 21 major coronary intervention centers in Korea, a total of 3,000 patients (anticipated) will be enrolled in this database between January 2010 and December 2014.

The aim of the study was to investigate long-term clinical results and predictors of adverse outcomes after percutaneous coronary intervention with 2nd generation drug-eluting stents for coronary bifurcation lesions in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Age >=19 years
* Any type of de novo bifurcation lesion in major epicardial artery: unprotected left main coronary bifurcation lesion, LAD - diagonal, LCX-OM, distal RCA bifurcation. (Excluding RCA-RV branch bifurcation, branch bifurcation)
* Side branch or LCX reference diameter >= 2.3 mm and at least stentable with 2.5 mm stent
* Treated with drug-eluting stent during the period of 2010. 1 ~ 2014. 12

Exclusion Criteria:

* Protected left main disease previous CABG for LAD or LCX territory
* Cardiogenic Shock
* History of CPR in the same hospitalization
* Patients with severe left ventricular systolic dysfunction (ejection fraction < 30%)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary bifurcation lesion treated with 2nd generation drug-eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 2648 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 5 years
  composite of cardiac death, myocardial infarction, or target lesion revascularization

SECONDARY OUTCOMES:
Cardiac death | 5 years
  All deaths were considered cardiac cause unless obvious non-cardiac causes could be identified
Myocardial infarction | 5 years
  an elevation of creatine kinase-myocardial band or troponin level greater than the upper limit of normal with concomitant ischemic symptoms or electrocardiography findings indicative of ischemia
Target lesion revascularization | 3 years
  repeat PCI of the lesion within 5 mm of the inserted stent
Stent thrombosis | 5 years
  the Academic Research Consortium as definite, probable, or possible

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi KH, Nam CW, Bruno F, Cho YK, De Luca L, Kang J, Mattesini A, Song YB, Truffa A, Kim HS, Wanha W, Chun WJ, Gili S, Helft G, Han SH, Cortese B, Lee CH, Escaned J, Yoon HJ, Chieffo A, Hahn JY, Gallone G, Choi SH, De Ferrari G, Koo BK, Quadri G, Hur SH, D'Ascenzo F, Gwon HC, de Filippo O. Differential Prognosis of True Bifurcation Lesions According to Left Main Versus Non-Left Main Location and Treatment Strategy. J Am Heart Assoc. 2025 Feb 4;14(3):e037657. doi: 10.1161/JAHA.124.037657. Epub 2025 Feb 3. PMID 39895551
- [Derived] Ahn HJ, Bruno F, Kang J, Hwang D, Yang HM, Han JK, De Luca L, de Filippo O, Mattesini A, Park KW, Truffa A, Wanha W, Song YB, Gili S, Chun WJ, Helft G, Hur SH, Cortese B, Han SH, Escaned J, Chieffo A, Choi KH, Gallone G, Doh JH, De Ferrari G, Hong SJ, Quadri G, Nam CW, Gwon HC, Kim HS, D'Ascenzo F, Koo BK. Sex Differences in Procedural Characteristics and Clinical Outcomes Among Patients Undergoing Bifurcation PCI. Korean Circ J. 2025 Jan;55(1):5-16. doi: 10.4070/kcj.2024.0172. Epub 2024 Oct 11. PMID 39601395
- [Derived] Lee JH, Youn YJ, Jeon HS, Lee JW, Ahn SG, Yoon J, Gwon HC, Song YB, Choi KH, Kim HS, Chun WJ, Hur SH, Nam CW, Cho YK, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Lim DS, Park JS, Hong MK, Doh JH, Cha KS, Kim DI, Lee SY, Chang K, Hwang BH, Choi SY, Jeong MH, Lee HJ. Transradial Versus Transfemoral Access for Bifurcation Percutaneous Coronary Intervention Using Second-Generation Drug-Eluting Stent. J Korean Med Sci. 2024 Mar 18;39(10):e111. doi: 10.3346/jkms.2024.39.e111. PMID 38501187
- [Derived] Choi KH, Bruno F, Cho YK, De Luca L, Song YB, Kang J, Mattesini A, Gwon HC, Truffa A, Kim HS, Wanha W, Chun WJ, Gili S, Hur SH, Helft G, Han SH, Cortese B, Lee CH, Escaned J, Yoon HJ, Chieffo A, Hahn JY, Gallone G, Choi SH, De Ferrari G, Koo BK, Quadri G, D'Ascenzo F, Nam CW, de Filippo O. Comparison of Outcomes Between 1- and 2-Stent Techniques for Medina Classification 0.0.1 Coronary Bifurcation Lesions. JACC Cardiovasc Interv. 2023 Sep 11;16(17):2083-2093. doi: 10.1016/j.jcin.2023.06.013. Epub 2023 Aug 9. PMID 37565964
- [Derived] Cha JJ, Hong SJ, Kim JH, Lim S, Joo HJ, Park JH, Yu CW, Kang J, Kim HS, Gwon HC, Chun WJ, Hur SH, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Yoon J, Park JS, Hong MK, Doh JH, Cha KS, Kim DI, Lee SY, Chang K, Hwang BH, Choi SY, Jeong MH, Song YB, Choi KH, Nam CW, Koo BK, Lim DS. Bifurcation strategies using second-generation drug-eluting stents on clinical outcomes in diabetic patients. Front Cardiovasc Med. 2022 Dec 21;9:1018802. doi: 10.3389/fcvm.2022.1018802. eCollection 2022. PMID 36620646
- [Derived] Lee CH, Nam CW, Cho YK, Yoon HJ, Kim KB, Gwon HC, Kim HS, Chun WJ, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Yoon J, Lim DS, Park JS, Hong MK, Lee SY, Cha KS, Kim DI, Bae JW, Chang K, Hwang BH, Choi SY, Jeong MH, Choi KH, Song YB, Hong SJ, Doh JH, Koo BK, Hur SH. 5-Year Outcome of Simple Crossover Stenting in Coronary Bifurcation Lesions Compared With Side Branch Opening. JACC Asia. 2021 Jun 15;1(1):53-64. doi: 10.1016/j.jacasi.2021.04.002. eCollection 2021 Jun. PMID 36338374
- [Derived] Choi KH, Song YB, Lee JM, Park TK, Yang JH, Hahn JY, Choi JH, Choi SH, Kim HS, Chun WJ, Hur SH, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Yoon J, Lim DS, Park JS, Hong MK, Doh JH, Cha KS, Kim DI, Lee SY, Chang K, Hwang BH, Choi SY, Jeong MH, Hong SJ, Nam CW, Koo BK, Gwon HC. Differential Long-Term Effects of First- and Second-Generation DES in Patients With Bifurcation Lesions Undergoing PCI. JACC Asia. 2021 Jun 15;1(1):68-79. doi: 10.1016/j.jacasi.2021.04.006. eCollection 2021 Jun. PMID 36338362
- [Derived] Lee JM, Lee SH, Kim J, Choi KH, Park TK, Yang JH, Song YB, Hahn JY, Choi JH, Choi SH, Kim HS, Chun WJ, Nam CW, Hur SH, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Yoon J, Lim DS, Park JS, Hong MK, Doh JH, Cha KS, Kim DI, Lee SY, Chang K, Hwang BH, Choi SY, Jeong MH, Hong SJ, Koo BK, Gwon HC. Ten-Year Trends in Coronary Bifurcation Percutaneous Coronary Intervention: Prognostic Effects of Patient and Lesion Characteristics, Devices, and Techniques. J Am Heart Assoc. 2021 Sep 21;10(18):e021632. doi: 10.1161/JAHA.121.021632. Epub 2021 Sep 13. PMID 34514841
- [Derived] Choi KH, Song YB, Lee JM, Park TK, Yang JH, Hahn JY, Choi JH, Choi SH, Kim HS, Chun WJ, Hur SH, Han SH, Rha SW, Chae IH, Jeong JO, Heo JH, Yoon J, Lim DS, Park JS, Hong MK, Doh JH, Cha KS, Kim DI, Lee SY, Chang K, Hwang BH, Choi SY, Jeong MH, Hong SJ, Nam CW, Koo BK, Gwon HC. Prognostic Effects of Treatment Strategies for Left Main Versus Non-Left Main Bifurcation Percutaneous Coronary Intervention With Current-Generation Drug-Eluting Stent. Circ Cardiovasc Interv. 2020 Feb;13(2):e008543. doi: 10.1161/CIRCINTERVENTIONS.119.008543. Epub 2020 Feb 7. PMID 32069106